CLINICAL TRIAL: NCT01066728
Title: CO2 Inhalation as a New Treatment Modality for Apnea of Prematurity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Children's Hospital Foundation of Manitoba (Unknown)
Responsible Party: Ruben E. Alvaro, MD, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E98:242
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-01

CONDITIONS: Apnea of Prematurity
Keywords: apnea; premature; infant; prematurity
MeSH Terms: conditions — Apnea; Premature Birth | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theophylline (Active Comparator): Oral loading dose of 6 mg per kilogram of body weight of theophylline followed by a maintenance dose of 2 mg per kilogram every 8 hours plus room air by nasal prongs at 0.5 l/min for 3 days.
  Interventions: Drug: Theophylline
- CO2 inhalation (Experimental): Equivalent loading and maintenance volume of oral normal saline plus CO2 (3% at the source, approximately 1% inhaled) with room air by nasal prongs at 0.5 l/min for 3 days
  Interventions: Other: CO2 inhalation

INTERVENTIONS:
Other: CO2 inhalation — Inhalation of CO2 (3% at the source, approximately 1% inhaled) with room air by nasal prongs at 0.5 l/min for 3 days
  Arms: CO2 inhalation
Drug: Theophylline
  Arms: Theophylline

SUMMARY:
The objective of the present proposed study is to discover whether, in the nursery setting, administration of low concentration inhaled CO2 (0.8%) for a prolonged period (3 days) can make breathing more regular with less apneic time than that observed with administration of theophylline. The hypothesis to be tested is that inhalation of low concentration CO2 (0.8%) will reduce apnea more effectively and will have fewer adverse side effects than theophylline.

DETAILED DESCRIPTION:
1. To discover whether, in the nursery setting, continuous administration of a low concentration of inhaled CO2 (0.8%) for a prolonged period (3 days) can make breathing in preterm infants more regular with less apneic time than that observed with theophylline.
2. To discover whether inhalation of low CO2 decreases apneas, particularly prolonged apneas (>20 seconds), more effectively than theophylline.
3. To discover whether short term (during hospitalization) and long term (2 years) adverse side effects are less pronounced with CO2 than with theophylline.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 27 and 32 weeks gestational age hospitalized in the neonatal intensive or intermediate care units
* Significant apnea, defined as 5 or more self-resolved apneas, or 2 or more apneas requiring intervention over a 12 hr period

Exclusion Criteria:

* Already on methylxanthine treatment
* On supplemental oxygen, nasal continuous positive airway pressure (CPAP)
* Had major congenital anomalies, sepsis, or other known causes of apnea

Ages: 27 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2001-08; Primary Completion 2005-09 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The decrease in total apnea time (duration of all apneic pauses ≥ 5 seconds) during administration of theophylline and carbon dioxide. | 3 days

SECONDARY OUTCOMES:
Decrease in the rate of long apneas (≥ 20 seconds) and the incidence of short term side effects | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Ruben E Alvaro, MD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - St Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba

REFERENCES:
- [Background] Al-Saif S, Alvaro R, Manfreda J, Kwiatkowski K, Cates D, Qurashi M, Rigatto H. A randomized controlled trial of theophylline versus CO2 inhalation for treating apnea of prematurity. J Pediatr. 2008 Oct;153(4):513-8. doi: 10.1016/j.jpeds.2008.04.025. Epub 2008 Jun 4. PMID 18534618
- [Background] Al-Aif S, Alvaro R, Manfreda J, Kwiatkowski K, Cates D, Rigatto H. Inhalation of low (0.5%-1.5%) CO2 as a potential treatment for apnea of prematurity. Semin Perinatol. 2001 Apr;25(2):100-6. doi: 10.1053/sper.2001.23199. PMID 11339662
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Long-term effects of caffeine therapy for apnea of prematurity. N Engl J Med. 2007 Nov 8;357(19):1893-902. doi: 10.1056/NEJMoa073679. PMID 17989382
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748
- [Background] Bucher HU, Duc G. Does caffeine prevent hypoxaemic episodes in premature infants? A randomized controlled trial. Eur J Pediatr. 1988 Apr;147(3):288-91. doi: 10.1007/BF00442697. PMID 3292249
- [Background] Dunwiddie TV, Masino SA. The role and regulation of adenosine in the central nervous system. Annu Rev Neurosci. 2001;24:31-55. doi: 10.1146/annurev.neuro.24.1.31. PMID 11283304
- [Background] Xie A, Rankin F, Rutherford R, Bradley TD. Effects of inhaled CO2 and added dead space on idiopathic central sleep apnea. J Appl Physiol (1985). 1997 Mar;82(3):918-26. doi: 10.1152/jappl.1997.82.3.918. PMID 9074983